CLINICAL TRIAL: NCT05578820
Title: An Open Multicenter Study of the Safety, Tolerability, and Pharmacokinetics of Different Doses of Stimotimagene Copolymerplasmid at Patients With Advanced-stage Solid Tumors With Cymeven® (Ganciclovir) Infusions
Brief Title: Safety, Tolerability and Pharmacokinetics Investigation of Stimotimagene Copolymerplasmid
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gene Surgery LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NTI1GSA
Record Dates: First submitted 2022-10-03; First posted 2022-10-13 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Sarcoma; Melanoma; Squamous Cell Carcinoma of Head and Neck; Breast Neoplasms; Uterine Cervical Neoplasms; Vulvar Neoplasms; Penile Neoplasms; Anus Neoplasms
MeSH Terms: conditions — Sarcoma; Melanoma; Squamous Cell Carcinoma of Head and Neck; Breast Neoplasms; Uterine Cervical Neoplasms; Vulvar Neoplasms; Penile Neoplasms; Anus Neoplasms | interventions — Ganciclovir

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose escalation phase (Experimental): Stimotimagene copolymerplasmid will be administered intratumoral once in a dose of 20 mkg of DNA per 1 cm3 of tumor (for cohort 1) and 40 mkg of DNA per 1 cm3 of tumor (for cohort 2).
  Ganciclovir (Cimeven®) will be administrated intravenous twice a day at 12-hour intervals for 15 days.
  Interventions: Biological: Stimotimagene copolymerplasmid; Drug: Ganciclovir
- Two times administration of Stimotimagene copolymerplasmid (Experimental): Stimotimagene copolymerplasmid will be administered intratumorally twice with 5-day interval in the optimal dose selected at previous stage of the trial.
  Ganciclovir (Cimeven®) will be administrated intravenous twice a day at 12-hour intervals for 15 days.
  Interventions: Biological: Stimotimagene copolymerplasmid; Drug: Ganciclovir
- Tree times administration of Stimotimagene copolymerplasmid (Experimental): Stimotimagene copolymerplasmid will be administered intratumorally three times with 5-day interval in the optimal dose selected at first stage of the trial.
  Ganciclovir (Cimeven®) will be administrated intravenous twice a day at 12-hour intervals for 15 days.
  Interventions: Biological: Stimotimagene copolymerplasmid; Drug: Ganciclovir

INTERVENTIONS:
Biological: Stimotimagene copolymerplasmid — Gene therapy drug, Intratumoral administration
  Other Names: AntioncoRAN-M
Drug: Ganciclovir — Antiviral drug, Intravenous administration
  Other Names: Cymeven®

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of different doses and administration regimens of Stimotimagene copolymerplasmid in patients with histologically confirmed diagnosis of solid tumor and/or its metastases.

DETAILED DESCRIPTION:
Stimotimagene copolymerplasmid is an anti-tumor gene therapy drug, contains super-coiled plasmid DNA encapsulated in polycationic envelope (PPT: polyethyleneimine (PEI) - polyethylene glycol (PEG) - TAT peptide). The plasmid encodes two therapeutic genes: herpes simplex virus thymidine kinase (HSVtk) and human granulocyte-macrophage colony-stimulating factor (hGM-CSF). HSVtk converts the prodrug ganciclovir to a toxin in cells that have been transfected by Stimotimagene copolymerplasmid, GM-CSF stimulates proliferation and differentiation of antigen-presenting cells.

Stimotimagene copolymerplasmid therapy is two-staged: (1) intratumoral injection of Stimotimagene copolymerplasmid, (2) intravenous administration of ganciclovir (Cimeven®) This is the first-in-human study of Stimotimagene copolymerplasmid which will be conducted in three arms. In this study dose escalation (Arm1) and number of drug administrations (Arms 2 and 3) will be explored. All study parts will investigate the safety, tolerability and pharmacokinetic profile of Stimotimagene copolymerplasmid.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18-75;
2. Histologically confirmed diagnosis of a solid tumor and/or its metastases: Sarcoma, Melanoma, Squamous Cell Carcinoma of Head and Neck, Breast Neoplasms, Uterine Cervical Neoplasms, Vulvar Neoplasms, Penile Neoplasms, Anus Neoplasms
3. Patients for whom surgery is not indicated;
4. Patients with exhausted methods of drug and radiation therapy;
5. Presence of clearly detectable and measurable by instrumental methods (ultrasound) tumor mass with a maximum size of at least 10 mm, palpable and accessible for intratumoral injection;
6. The injected with the test drug tumor mass must not be located near large blood vessels or nerves;
7. General health according to the ECOG scale 0-2;
8. Life expectancy of at least 3 months;
9. Hemoglobin ≥ 90 g/l;
10. Absolute neutrophil count ≥ 1500/mm3;
11. Platelet count ≥ 100,000/mm3;
12. Creatinine clearance ≥ 70 ml/min;
13. Quick Prothrombin Time more than 55%;
14. At least 4 weeks or at least 5 elimination half-lives must elapse between previous chemotherapy, targeted therapy, radiotherapy, immunotherapy, or experimental antitumor therapy and administration of the study drug;
15. Patients must recover from any previous surgery, radiotherapy, localized therapy, or systemic therapy to grade 1 or lower adverse reactions (except alopecia or anemia, for which grade 2 is acceptable);
16. Women of childbearing age (not menopausal or surgically sterilized) and men who are sexually active should use a reliable method of contraception (acceptable methods of contraception in this study are: IUDs, oral contraceptives, contraceptive patch, long-acting injectable contraceptives, dual barrier method (condom and spermicide, diaphragm and spermicide) during the study and at least 30 days after the last dose of Cymeven® for female patients and at least 90 days after the last dose of Cymeven® for male patients;
17. Ability to follow protocol procedures throughout the study;
18. Presence of Patient Informed Consent to Participate in a Clinical Trial.

Exclusion Criteria:

1. The investigator's concern that injecting the drug into the tumor mass may lead to life-threatening side effects, if tumor swelling or inflammation occurs after treatment;
2. History of hypersensitivity to ganciclovir, valganciclovir, or any other component of Cymeven®;
3. History of hypersensitivity to acyclovir or pencyclovir (or their prodrugs valacyclovir or famciclovir, respectively);
4. History of allergic reactions to antibiotics;
5. History of allergic reaction to polyethylene glycol or polyethyleneimine;
6. The following medications are scheduled to be taken during the potential therapy period:

   * imipenem/cylastatin
   * drugs that have myelosuppressive effects or impair renal function: nucleoside analogues (e.g., zidovudine, didanosine, stavudine), immunosuppressants (e.g., cyclosporine, tacrolimus, mycophenolate mofetil), anticancer drugs (e.g, doxorubicin, vincristine, vinblastine, hydroxyurea) and anti-infective drugs (e.g., trimethoprim/sulfamides, dapsone, amphotericin B, flucytosine, pentamidine);
   * probenecid;
7. Pregnancy or lactation;
8. Presence of primary multiple malignant diseases;
9. Presence of connection of the tumor mass with the main vessels according to ultrasound/CT/MRI data;
10. Radiation damage (ulceration, necrosis);
11. High risk/continued bleeding;
12. Systemic connective tissue disease (scleroderma, etc.);
13. Exacerbation of allergic diseases at the time of inclusion in the study;
14. Liver function disorder;
15. Presence of acute and acute chronic infections within the last 4 weeks before inclusion in the study (including tuberculosis, abscess, phlegmon);
16. Exacerbations of chronic diseases of the cardiovascular, bronchopulmonary, urogenital, gastrointestinal, musculoskeletal, nervous and immune systems at the time of inclusion in the study;
17. Presence of mental illness;
18. A history of active primary immunodeficiency;
19. Presence of HIV, active hepatitis B or C;
20. Brain metastases, carcinomatous meningitis at the moment of inclusion in the study;
21. Patient's participation in another clinical trial less than 30 days before inclusion in this study;
22. Any condition that, in the opinion of the investigator, might interfere with adequate treatment delivery, including difficult contact with the patient (inadequate perception of information provided about the patient's condition and planned/conducted treatment, refusal to comply with recommendations).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-04-11 (Actual)

PRIMARY OUTCOMES:
Safety (Presence/absence of dose-limiting toxicities (DLTs)) | Through study completion, an average of 1 year
  Assessment of presence/absence of dose-limiting toxicities (DLTs)
Safety (Frequency and severity of adverse events (CTCAE classification)) | Through study completion, an average of 1 year
  Assessment of frequency and severity of adverse events (CTCAE classification)
Safety (Number of cases of early termination of participation in the study due to the development of Serious Adverse Events and Other Adverse Events associated with the study therapy) | Through study completion, an average of 1 year
  Assessment of number of cases of early termination of participation in the study due to the development of Serious Adverse Events and Other Adverse Events associated with the study therapy)
Pharmacokinetics (Quantitative content of plasmid DNA (pTKhGM) in patients' peripheral blood) | Through study completion, an average of 1 year
  Assessment of quantitative content of plasmid DNA (pTKhGM) in patients' peripheral blood at:
  Day -1 (baseline), Day 1 (4 h and 8 h after drug administration), Day 2 (24 h after drug administration), Day 3 (48 h after drug administration), Days 5, 7, 12, 17, 25, 30±3, 60±5, 90±7, 130±3 for patients from 1st step of the study; Day -1 (baseline), Day 1 (4 h and 8 h after drug administration), Day 2 (24 h after drug administration), Day 3 (48 h after drug administration), Day 6 (before drug administration and 8 h after drug administration), Days 7, 12, 17, 25, 30±3, 60±5, 90±7, 130±3 for patients from 2nd step of the study; Day -1 (baseline), Day 1 (4 h and 8 h after drug administration), Day 2 (24 h after drug administration), Day 3 (48 h after drug administration), Day 6 (before drug administration and 8 h after drug administration), Day 7, Day 11 (before drug administration and 8 h after drug administration), Days 12, 17, 25, 30±3, 60±5, 90±7, 130±3 for patients from 3rd step of the
Pharmacokinetics (Quantitative content of plasmid DNA (pTKhGM) in patients' urine) | Through study completion, an average of 1 year
  Assessment of quantitative content of plasmid DNA (pTKhGM) in patients' urine at:
  Day -1 (baseline), Day 1 (4 h and 8 h after drug administration), Day 2 (24 h after drug administration), Day 3 (48 h after drug administration), Days 5, 7, 12, 17, 25, 30±3, 60±5, 90±7, 130±3 for patients from 1st step of the study; Day -1 (baseline), Day 1 (4 h and 8 h after drug administration), Day 2 (24 h after drug administration), Day 3 (48 h after drug administration), Day 6 (before drug administration and 8 h after drug administration), Days 7, 12, 17, 25, 30±3, 60±5, 90±7, 130±3 for patients from 2nd step of the study; Day -1 (baseline), Day 1 (4 h and 8 h after drug administration), Day 2 (24 h after drug administration), Day 3 (48 h after drug administration), Day 6 (before drug administration and 8 h after drug administration), Day 7, Day 11 (before drug administration and 8 h after drug administration), Days 12, 17, 25, 30±3, 60±5, 90±7, 130±3 for patients from 3rd step of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Irina Alekseenko, Study Director
Locations (4):
- Russia (4):
  - GBUZ Moscow Clinical Scientific Center named after Loginov MHD, Moscow
  - FSBI N.N. Blokhin National Medical Research Center of Oncology of the Ministry of Health of Russia, Moscow
  - FSBI National Medical Research Center for Obstetrics, Gynecology and Perinatology named after Academician V.I.Kulakov of the Ministry of Health of Russia, Moscow
  - National Medical Research Radiological Centre of the Ministry of Health of the Russian Federation, Moscow